CLINICAL TRIAL: NCT01741844
Title: Regulatory Post Marketing Surveillance of Intelence Tablet
Brief Title: A Post Marketing Survey Study to Evaluate the Safety and Effectiveness of Intelence
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100806; TMC125HIV4017 (Other: Janssen Korea, Ltd., Korea); Intelene PMS (Other: Janssen Korea, Ltd., Korea); ETR-C-11-KR-001-V04 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Acquired Immune Deficiency Syndrome
Keywords: Acquired Immune Deficiency Syndrome; TMC125; Etravirine; Intelence; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Etravirine: Patients having Acquired Immune Deficiency Syndrome (AIDS) will be taking etravirine as per recommended doses.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Etravirine 200 mg will be adminstered twice daily in patients with Acquired Immune Deficiency Syndrome (AIDS).

SUMMARY:
The purpose of this study is to assess the safety data of etravirine in a natural clinical practice.

DETAILED DESCRIPTION:
This is a non-interventional (a scientific study to make a clear and easy understanding of the cause and effect relationship), prospective (in which the participants are first identified and then followed forward as time passes), consecutive survey for collecting safety and efficacy data of etravirine in treatment of Acquired Immune Deficiency Syndrome (AIDS) in a natural clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are prescribed with etravirine for treatment of Acquired Immune Deficiency Syndrome (AIDS)

Exclusion Criteria:

* Known hypersensitivity to Intelence
* Intelence coadministered with medicinal products that are highly dependent on CYP3A and CYP2C9 for clearance
* Patients with galactose intoralance, Lapp lactase deficiency, and glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who are diagnosed with Acquired Immune Deficiency Syndrome (AIDS), and who are prescribed with etravirine for treatment of AIDS.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 30 days from end of treatment

SECONDARY OUTCOMES:
Number of patients with viral load | Screening, Week 12, Week 24
Number of patients with CD4 T-cell count | Screening, Week 12, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (1):
- Daegu, South Korea